CLINICAL TRIAL: NCT05538481
Title: A Prospective Study to Identify and Measure the Cultural Values and Palliative Care Preferences of Hindu Patients With Cancer and Their Caregivers
Brief Title: Study to Identify and Measure the Values and Palliative Care Pref. of Hindu Patients and Their Caregivers
Status: Withdrawn | Type: Observational
Why Stopped: Sponsor Investigator transferred from institution
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Atrium Health Levine Cancer Institute (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00085986; LCI-SUPP-NOS-HCV-001 (Other: Levine Cancer Institute)
Record Dates: First submitted 2022-09-05; First posted 2022-09-13 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-07

CONDITIONS: Neoplasms
Keywords: Palliative Care; Hindu Culture; Community-based Participatory Research
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Focus Group: A total of 16 participants, including patients and caregivers, will be enrolled for 2 focus groups (group of 8 patients with cancer and group of 8 caregivers).
  Interventions: Other: Semi-structured interview; Other: Systems of Belief Inventory (SBI-15R)
- Cognitive Interviews Group: A total of up to 30 participants will be enrolled in this cohort, and up to 3 rounds of cognitive interviews will be conducted. This cohort of participants will be enrolled after survey development based on the themes identified from the focus group analyses.
  Interventions: Other: Developed survey completion; Other: Systems of Belief Inventory (SBI-15R)

INTERVENTIONS:
Other: Semi-structured interview — A collection of individual cultural values and palliative care preferences within the focus group meetings
  Groups: Focus Group
Other: Developed survey completion — A collection of individual responses to a survey created after focus group completion and analysis
  Groups: Cognitive Interviews Group
Other: Systems of Belief Inventory (SBI-15R) — A 15-item questionnaire designed to measure religious and spiritual beliefs and practices and the social support derived from a community sharing those beliefs.

SUMMARY:
Historically, palliative care in the US has been rooted in the cultural values of a Caucasian, Christian middle class. Greater understanding of how culture influences the delivery of palliative care to minority patients is needed to achieve health equity.

The purpose of this study is to learn more about the cultural values (Hindu customs and beliefs) and palliative care (specialized care for people living with a serious illness) preferences of the Hindu community. To the study team's knowledge, there has not been another study that has used a research approach to help better understand and measure the cultural values and palliative care preferences of Hindu participants with cancer and their caregivers.

DETAILED DESCRIPTION:
This is a cross-sectional study of Hindu patients with cancer in Charlotte and surrounding areas and their Hindu caregivers. This study will use the methods and principles of Community-based participatory research (CBPR).

Before enrollment of participants, a Community Advisory Group (CAG) will be formed, which represents the Hindu community's perspective in the research project and facilitates interactions with Hindu patients with cancer and caregivers. The CAG will be composed of 8-10 members, including healthcare professionals, leaders, patients with cancer, and their caregivers - identified by members from three Hindu institutions, Bochasanwasi Shri Akshar Purushottam Swaminarayan Sanstha (BAPS), Hindu Center of Charlotte, and Trimurti Temple Devasthanam, in Charlotte and surrounding areas. Charlotte is one of the two areas in NC with the fastest growing Indian population. The role of the CAG is to provide input throughout both parts of the study.

There will be two cohorts of patients with cancer/caregivers: 1) focus group cohort and 2) cognitive interview cohort. Data about cultural values and palliative care preferences collected from focus group participants (Cohort 1) will be analyzed using an inductive thematic analysis approach and will be used for survey development. The survey will be validated with cognitive interviews (Cohort 2). After any needed modifications, the final survey will be created and presented to all study participants. All of the study participants will also have the opportunity to review the survey to ensure that the questions reflect their real-world experiences. The investigators hypothesize that this final survey will be an effective tool to measure the cultural values and palliative care preferences of Hindu patients and their caregivers.

Participants will be enrolled over approximately 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Verbal informed consent by the patient or caregiver
2. Age ≥ 18 years at the time of consent
3. Participants must be a cancer patient or caregiver and/or:

   * Self-identified Hindu
   * Cancer patients must have received most of their cancer care in Charlotte and surrounding areas within the past 5 years from enrollment
   * Caregivers must be caring for a patient who meets the above criteria and is too ill to participate or cared for a cancer patient who met the above criteria but died within the past 5 years from enrollment
4. Ability to read, speak, and understand English
5. As determined by the enrolling investigator, the ability of the participant to understand and comply with study procedures for the entire length of the study

Exclusion Criteria:

1. Lack of access to the technology required to attend virtual meetings and complete study surveys electronically (e.g., internet in home setting)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with cancer ≥18 years of age and self-identified Hindus who received the majority of their cancer care in Charlotte and surrounding areas within the past 5 years will be identified by the investigators and Community Advisory Group members.
  Or
  Caregivers ≥18 years of age and self-identified Hindus who are caring for an eligible Hindu patient or cared for an eligible Hindu patient who died ≤ 5 years will be identified by the investigators and Community Advisory Group members.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-06 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
To identify the cultural values and palliative care preferences of Hindu patients with cancer and caregivers in Charlotte and surrounding areas. | approx. 12 months
  Qualitative analysis will occur on collected sociodemographic data and responses to Systems of Belief Investigator (SBI-15R). Using MAXQDA Analytics Pro software, themes will be identified for coding based on the repetition of specific words, phrases, and opinions, use of language and general thought patterns, as well as specific topics that dominated the focus group discussion. A theme will be defined as an issue raised or discussed by ≥2 members in that focus group. This phase of the study will conclude when new themes no longer emerge, i.e., thematic saturation is reached.
To develop and validate the content of a survey of Hindu cultural values and palliative care preferences to measure their prevalence in a larger cohort. | approx. 12 months
  Qualitative analysis will be performed based on Cognitive interviews utilizing created survey. Items that have <3 instances of being identified by participants as being problematic will be retained and will not be retested in any subsequent cognitive interview rounds. If any aspect of the measure has ≥3 instances of being identified by the participant as being problematic in the final round, that aspect will be removed from the final survey.

CONTACTS AND LOCATIONS:
Overall Officials: Rushil Patel, MD, Principal Investigator — Atrium Health Levine Cancer Institute
Locations (1):
- Levine Cancer Institute, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No